CLINICAL TRIAL: NCT07281989
Title: Sound Stops Stress Study: Evaluating the WAVwatch Effect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 37459
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single arm where participants act as their own control
  Interventions: Device: WAVWatch 2.0

INTERVENTIONS:
Device: WAVWatch 2.0 — The WAVwatch 2.0, a wrist-worn device intervention, leverages 'calming' frequencies to reduce stress and non-clinically relevant anxiety, aligning with scientific evidence supporting sound therapy's potential.

SUMMARY:
Sound Off Stress Study seeks to discover if WAVwatch 2.0-a sleek, wearable sound frequency device-can support mental harmony.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to rigorously evaluate the efficacy of the WAVwatch 2.0, a cutting-edge sound frequency device, in mitigating stress and everyday anxiety. In an era where stress pervades our daily lives, the need for innovative, science-backed solutions has never been more critical. Amidst the growing social media enthusiasm surrounding sound therapy's tranquil effects, this study seeks to scientifically substantiate the capabilities of WAVwatch 2.0, aiming to either validate or debunk the widespread claims of its beneficial impact on mental states.

The primary objective is to equip participants with precise, data-driven insights regarding the potential of WAVwatch 2.0 to diminish stress and anxiety levels. By partaking in this investigation, individuals will gain a personal understanding of their mental wellness journey, assessing firsthand whether this sophisticated, wearable technology can integrate seamlessly into their lives and foster the tranquility and equilibrium they aspire to achieve.

The core aims and objectives of this trial center around the thorough assessment of WAVwatch 2.0's effectiveness in lowering stress and anxiety, whilst concurrently promoting overall life satisfaction. Through personalized feedback, participants will be endowed with the knowledge necessary to make enlightened decisions regarding their stress management strategies and potential financial commitments to wellness technologies.

The significance and impact of this study are vast, with the potential to transform the landscape of personal stress management. By delivering evidence-based insights into the efficacy of sound frequency technology in enhancing mental wellness, this research could pave the way for more informed, individualized choices in non-clinical anxiety relief methods. While WAVwatch 2.0 may not be universally applicable, its evaluation serves as a critical step towards diversifying and enriching the arsenal of tools available for achieving mental well-being, thus empowering participants to make well-informed decisions concerning their wellness journeys.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Exclusion Criteria:

* Individuals with skin sensitivities
* Individuals with auditory conditions
* Individuals with severe anxiety or mental health disorders
* Pregnancy
* Individuals prone to irritation or frustration

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (Past Week Version) | Change from baseline (Day 1-3) in perceived stress levels at 4 weeks after the start of the intervention (Day 27-33)
  The Perceived Stress Scale (Past Week Version) is a modified version of the classic stress assessment tool that evaluates stress levels based on recent experiences within the last week. This scale helps in understanding how various situations have recently affected an individual's feelings and perceived stress levels. By focusing on a shorter time frame, it provides a more immediate assessment of stress, which can be particularly useful for quickly evaluating the effectiveness of stress management strategies or interventions. The tool retains its original structure, ensuring its reliability while making it more relevant for current stress evaluation.
General Anxiety Disorder (GAD-7) | Change from baseline (Day 1-3) in anxiety severity at 4 weeks after the start of the intervention (Day 27-33)
  The GAD-7 is a 7-item questionnaire used to assess the severity of generalized anxiety disorder (GAD) in adults. The score is based on the responses to seven questions about the frequency of common anxiety symptoms over the past two weeks.
NIH Toolbox® Item Bank v3.0 - General Life Satisfaction (Ages 18+) | Change from baseline (Day 1-3) in general life satisfaction at 4 weeks after the start of the intervention (Day 27-33)
  This is a survey aimed at assessing the general life satisfaction of individuals aged 18 and above. Participants are asked a series of questions to which they can respond by indicating their level of agreement or disagreement.
Depression, Anxiety and Stress Scales (DASS-21) Survey | Change from baseline (Day 1-3) in depression, anxiety, and stress levels at 4 weeks after the start of the intervention (Day 27-33)
  The Depression, Anxiety, and Stress Scales (DASS-21) is a widely recognized psychological assessment tool designed to measure the severity of symptoms related to depression, anxiety, and stress. It consists of 21 questions that assess various emotional and psychological factors. Participants are asked to rate the frequency and intensity of their experiences over the past week. The DASS-21 survey provides a quick and reliable way for clinicians, researchers, and individuals to gauge their levels of depression, anxiety, and stress, making it a valuable instrument for mental health assessment and research.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=37454